CLINICAL TRIAL: NCT02302547
Title: Randomized Clinical Trial to Evaluate the Interest of a Down-scaled Treatment Strategy Using Dual Therapy (Nucleoside Analogs) in HIV Infected Patients Already Being Treated Using Triple Therapy, Who Present With a Successful Virological Control and for Which the HIV Reservoir is Low to Moderate
Brief Title: Trial to Evaluate the Interest of a Reductive Anti Retroviral Strategy Using Dual Therapy Inspite of Triple Therapy
Acronym: TRULIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: HOSPITAL, ORLEANS (Unknown); Poitiers University Hospital (Other); Centre Hospitalier de La Rochelle (Other); HOSPITAL, SAINTES (Unknown); HOSPITAL, FOCH (Unknown); HOSPITAL, CAEN (Unknown); Henri Mondor University Hospital (Other); HOSPITAL, HOTEL DIEU (Unknown); HOSPITAL, CHARTRES (Unknown); HOSPITAL, SAINT LOUIS (Unknown); Tourcoing Hospital (Other); Central Hospital, NIORT (Unknown); Tenon Hospital, Paris (Other); Central Hospital, Nancy, France (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHAO13-TP/TRULIGHT
Record Dates: First submitted 2014-10-14; First posted 2014-11-27 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2018-11

CONDITIONS: HIV
Keywords: HIV-DNA; dual therapy; NRTI; virological control; truvada®
MeSH Terms: interventions — Nevirapine; etravirine; Rilpivirine; Indinavir; fosamprenavir; tipranavir; Darunavir; Atazanavir Sulfate; Lopinavir; dolutegravir; Dual Anti-Platelet Therapy; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triple therapy (Active Comparator): Tenofovir Disoproxil Fumarate (nucleotide reverse transcriptase inhibitor) + Emtricitabine (nucleoside reverse transcriptase inhibitor) + third agent (boosted protease inhibitor or unboosted protease inhibitor or integrase inhibitor or celsentri or non-nucleoside reverse transcriptase inhibitor).
  Interventions: Drug: triple therapy
- dual therapy (Experimental): Truvada®"245mg":oral administration Tenofovir Disoproxil Fumarate (nucleotide reverse transcriptase inhibitor) + Emtricitabine (nucleoside reverse transcriptase inhibitor)
  Interventions: Drug: dual therapy

INTERVENTIONS:
Drug: triple therapy — Dosage treatment and usual prescription
  Other Names: Tenofovir+Emtricitabine+Third agent (Including a non nucleoside reverse transcriptase inhibitor: efavirenz or nevirapine or etravirine or rilpivirine; Tenofovir+Emtricitabine+Third agent (Including a ritonavir-boosted protease inhibitor : saquinavir or indinavir or fosamprenavir or tipranavir or darunavir or atazanavir or lopinavir; Tenofovir+Emtricitabine+Third agent (Including an unboosted protease inhibitor: atazanavir or indinavir; Tenofovir+Emtricitabine+Third agent (Including an integrase inhibitor raltegravir or dolutegravir or cobicistat-boosted elvitegravir; Tenofovir+Emtricitabine+Third agent (Including a fusion inhibitor: enfuvirtide or a CCR5 antagonist :maraviroc
  Arms: triple therapy
Drug: dual therapy — 1 tablet (200mg/245mg) daily for 48 weeks
  Other Names: Truvada®
  Arms: dual therapy

SUMMARY:
In the early 2000s, the "TRILEGE©" study was realized to determine if the reductive anti retroviral strategy from an initial triple therapy (based on a protease inhibitor as the third agent) towards a dual therapy of nucleoside analogs (in particular the association of "zidovudine +lamivudine") for patients infected by HIV and stabilized for at least 3 months at a threshold value of 400 copies/ml, would allow to obtain a well-controlled plasmatic viral load, with an aim to reduce the long-term side effects of the treatment.

The afore mentioned study showed that the reductive anti retroviral strategy was a failure. No study has as yet to revaluate this strategy, in particular in the current context of antiretroviral treatments.

Indeed, modern nucleoside inhibitors (Kivexa®, Truvada®) have extended half-lives as well as a superior intrinsic power as compared to treatments proposed in the initial "TRILEGE©" study. Furthermore, the better quality of current triple therapy (as compared to that used 10 years ago) has lead to substantial viral reservoir reduction.

Currently, a small number of patients is being successfully treated in the long-term (viral load < 20 copies/ml) using nucleoside analog dual therapy. The particular characteristics of these patients have yet to be thoroughly investigated.

The patients concerned were all treated prematurely before ever passing below 200 lymphocytes T CD4/mm3. It occurred that all these patients presented a low viral reservoir as measured by HIV DNA quantification (< 2,7 log copies/106 PBMC).

Therefore, by targeting patients who have (1) a strong immune restoration, (2) a low HIV DNA value and (3) a very good observance, the investigators emit the hypothesis that, reductive anti retroviral strategy that would consist in changing from a conventional triple therapy towards a Nucleoside reverse-transcriptase inhibitors dual therapy, could allow for durable control of viral replication with the concomitant benefice of reduced antiretroviral side effects and cost.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patient
* Initial TT ARV started above (or equal to) 150 / mm3 LT CD4, and 18 months prior to inclusion in the study
* Ongoing antiretroviral therapy combining tenofovir + emtricitabine + a 3rd agent (IP / r, IP, NNRTI, II, Inhibitors) with at least one undetectable viral load (CV <50 copies / mL) after introduction of the latter treatment.
* Patient in virological success: CV <50 copies / mL for at least 12 months, including visit to selection.
* Absence of previous therapeutic failure: no viral load ≥ 200 copies / mL (after 6 months of treatment) (Except in the case of a justified therapeutic interruption: travel, stock-out ...) and of obtaining success Virologic after introduction of treatment, without concept of genotypic resistance known to the ARVs used.
* Cellular DNA-HIV <2.7 log copies / 106 PBMC
* Zenith RNA-HIV <150,000 copies / ml (excluding viral load values during primary infection if it is documented)
* No genotypic resistance to currently used and known ARVs
* Patient who has given written informed consent
* Affiliate or beneficiary of a social security scheme
* Patient followed on an outpatient basis, age ≥ 18 years.

Exclusion Criteria:

* Non-compliant patient
* Subject is pregnant, or lactating, or of childbearing potential and without contraception
* Active opportunistic infections
* Major overweight (BMI ≥ 40)
* Severe renal pathology (creatinine clearance < 30ml/min)
* Cirrhosis or severe liver failure (factor V < 50%)
* Prognosis threatened within 6 months
* Circumstances that may impair judgment or understanding of the information given to the patient
* Malabsorption syndromes
* The following laboratory criteria:

  * Serum ASAT,ALAT > 5 x upper limit of normal (ULN)
  * Thrombocytopenia with platelet count < 50.000/ml
  * Anemia with hemoglobin < 8g/dl
  * Polynuclear neutrophil count < 500/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Viral Load at 48 weeks | 48 weeks
  Percentage of patient having a viral load < 50 copies/ml in each arm reductive anti retroviral strategy from an original backbone of 2 Nucleoside reverse transcriptase inhibitors (Tenofovir Disoproxil Fumarate+ Emtricitabine) coupled to a third agent, towards a therapeutic strategy containing the backbone therapy alone (Truvada®).

SECONDARY OUTCOMES:
Change from week 4 in Viral load at 48 weeks | between 4 weeks and 48 weeks
  percentage of patients having a viral load between 50 and 400 copies/ml between week 4 and week 48
CD 4 level in each arm | 48 weeks
  delta CD 4 measurement in each arm
Change from day 0 in HIV - DNA at week 48 | day 0 and 48 weeks
  HIV DNA evolution between day 0 and week 48 in each arm
RNA and DNA viral load (sub study) | Time Frame: Week 24 to Week 48
  RNA and DNA viral load in the genital tract (cervico-vaginal secretions or sperm): comparison between arms

CONTACTS AND LOCATIONS:
Overall Officials: LOUIS BERNARD, Pr, Principal Investigator — CHRU de TOURS; GWENAEL LE MOAL, Dr, Principal Investigator — Poitiers University Hospital; MARIAM RONCATO- SABERAN, Dr, Principal Investigator — CH de LA ROCHELLE; THIERRY PASDELOUPS, Dr, Principal Investigator — CH de SAINTES; DAVID ZUCMAN, Dr, Principal Investigator — HOPITAL de FOCH; RENAUD VERDON, Pr, Principal Investigator — University Hospital, Caen; SEBASTIEN GALLIEN, Pr, Principal Investigator — CHU d'HENRI MONDOR; JEAN - PAUL VIARD, Pr, Principal Investigator — CH d'HOTEL DIEU; MARC LESTELLE, Dr, Principal Investigator — CH de CHARTRES; JEAN - MICHEL MOLINA, Pr, Principal Investigator — CHU SAINT LOUIS; FAÏZA AJANA, Dr, Principal Investigator — CH de TOURCOING; SIMON SUNDER, Dr, Principal Investigator — CH de NIORT; Gilles PIALOUX, Pr, Principal Investigator — HOSPITAL TENON; Thierry MAY, Dr, Principal Investigator — Central Hospital, Nancy, France; Manuel ETIENNE, Dr, Principal Investigator — University Hospital, Rouen
Locations (16):
- France (16):
  - Unité des Maladies Infectieuses, CHU de CAEN, Caen
  - Service des Maladies Infectieuses, CHR Orléans La Source, ORLEANS CEDEX 2, CHR d'ORLEANS
  - Service d'Immunologie Clinique centre de Vaccination anti- VIH ANRS Hopital Henri- Mondor, Créteil
  - Service de Médecine Interne et Maladies Infectieuses, Groupe Hospitalier La Rochelle, Cedex 01, La Rochelle
  - Service de Pneumologie, centre Hospitalier Fontenoy, CH de CHARTRES, Le Coudray
  - CHU de NANCY, Nancy
  - Service des maladies Infectieuses et tropicales, CH GEORGES RENON, Niort
  - Service des Maladies Infectieuses et tropicales, APHP SAINT LOUIS, Paris
  - Hospital Tenon, Paris
  - Centre de diagnostic et thérapeutique, Hopital Hotel Dieu, Paris
  - Consultation Maladies Infectieuses, Chu de Poitiers, Cedex, Poitiers
  - Maladies Infectieuses, CHU de ROUEN, Rouen
  - Service de Médecine Interne, CH de SAINTONGE- BP 326, Saintes
  - Médecine Interne, Hôpital FOCH, Suresnes
  - Service Universitaire des Maladies Infectieuses et du Voyageur, CH DRON, Tourcoing
  - Service de Medecine Interne et Maladies Infectieuses, CHRU BRETONNEAU, TOURS CEDEX9, Tours

REFERENCES:
- [Background] Prazuck T, Verdon R, Le Moal G, Ajana F, Bernard L, Sunder S, Roncato-Saberan M, Ponscarme D, Etienne M, Viard JP, Pasdeloup T, Darasteanu I, Pialoux G, de la Blanchardiere A, Avettand-Fenoel V, Parienti JJ, Hocqueloux L; TRULIGHT Study Team. Tenofovir disoproxil fumarate and emtricitabine maintenance strategy in virologically controlled adults with low HIV-1 DNA: 48 week results from a randomized, open-label, non-inferiority trial. J Antimicrob Chemother. 2021 May 12;76(6):1564-1572. doi: 10.1093/jac/dkab038. PMID 33724373
- [Derived] Hocqueloux L, Gubavu C, Prazuck T, De Dieuleveult B, Guinard J, Seve A, Mille C, Gardiennet E, Lopez P, Rouzioux C, Lefeuvre S, Avettand-Fenoel V. Genital Human Immunodeficiency Virus-1 RNA and DNA Shedding in Virologically Suppressed Individuals Switching From Triple- to Dual- or Monotherapy: Pooled Results From 2 Randomized, Controlled Trials. Clin Infect Dis. 2020 Apr 15;70(9):1973-1979. doi: 10.1093/cid/ciz511. PMID 31350995